CLINICAL TRIAL: NCT04501367
Title: Assessing the Efficacy and Safety fo DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert(s) When Placed Within the Lower Eye Lid Canaliculus or Both the Upper and Lower Canaliculi for the Treatment of Pain, Inflammation, and Cystoid Macular Edema Following 27 Gauge Vitrectomy With Internal Limiting Membrane Peel for the Treatment of Retinal Edema Associated With Macular Pucker.
Brief Title: Assessing the Efficacy and Safety fo DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert(s) for the Treatment of Pain, Inflammation, and Cystoid Macular Edema Following 27 Gauge Vitrectomy With Internal Limiting Membrane Peel for the Treatment of Retinal Edema Associated With Macular Pucker.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kovach Eye Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kovacheye
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Vitrectomy; Macular Pucker; Retinal Edema
MeSH Terms: conditions — Epiretinal Membrane; Papilledema

STUDY DESIGN:
Intervention Model Description: In patients who undergo vitrectomy with internal limiting membrane peel surgery , subjects will be randomized to three groups and be followed for a period of two months. One group will be selected to receive one DEXTENZA (in the lower canaliculus), the second group will receive two DEXTENZA (upper and lower canaliculi) and the third group will receive prednisolone acetate 1% (control eye) . All groups will receive a subconjunctival dexamethasone injection at the time of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DEXTENZA Group (Experimental): Patients undergoing vitrectomy with internal limiting membrane peel
  Interventions: Drug: Dexamethasone Intracanalicular Insert, 0.4 mg
- Second DEXTENZA Group (Experimental): Patients undergoing vitrectomy with internal limiting membrane peel
  Interventions: Drug: Dexamethasone Intracanalicular Insert, 0.4 mg
- Topical Prednisolone Acetate 1% Group (Experimental): Patients undergoing vitrectomy with internal limiting membrane peel
  Interventions: Drug: Prednisone acetate 1%

INTERVENTIONS:
Drug: Dexamethasone Intracanalicular Insert, 0.4 mg — To determine post-surgical resolution of pain, inflammation, and cystoid macular edema outcomes when treated with one DEXTENZA (lower eye lid canaliculus) compared to topical steroid treatment in patients who undergo vitrectomy with internal limiting membrane peel surgery
  Arms: DEXTENZA Group
Drug: Dexamethasone Intracanalicular Insert, 0.4 mg — To determine post-surgical resolution of pain, inflammation, and cystoid macular edema outcomes when treated with two DEXTENZA (upper and lower canaliculi) compared to topical steroid treatment in patients who undergo vitrectomy with internal limiting membrane peel surgery
  Arms: Second DEXTENZA Group
Drug: Prednisone acetate 1% — To reduce post-surgical pain and inflammation in patients who undergo vitrectomy with internal limiting membrane peel surgery
  Arms: Topical Prednisolone Acetate 1% Group

SUMMARY:
Assessing the efficacy and safety of DEXTENZA, sustained release dexamethasone 0.4 mg inserts following 27 gauge vitrectomy with internal limiting membrane peel

DETAILED DESCRIPTION:
Assessing the efficacy and safety of DEXTENZA, sustained release dexamethasone 0.4 mg inserts, when placed within the lower eye lid canaliculus or both the upper and lower canaliculi for the treatment of pain, inflammation, and cystoid macular edema following 27 gauge vitrectomy with internal limiting membrane peel for the treatment of retinal edema associated with macular pucker

ELIGIBILITY:
Inclusion Criteria: A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Symptomatic macular pucker with retinal edema
* Age 18 years and older
* Scheduled vitrectomy and internal limiting membrane peel
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria: A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18
* Pregnancy ( must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye (s)
* Hypersensitivity to dexamethasone or prednisolone eye drops
* Patients being treated with immunomodulating agents in the study eye(s)
* Patient being treated with immunosuppressants and/or oral steroids
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in retina edema | assessed on day 30 and day 60
  As measured by Optical Coherence Tomography (OCT)

SECONDARY OUTCOMES:
Mean change in Inflammation ( Cell and Flare) | as assessed on days 1, 7, 30, 60
  As measured by SUN (Standardization of Uveitis Nomenclature) grading scale;absence of cell to be defined as a grade of 0-0.5 and absence of flare to be defined as a grade of 0-1
Mean change in pain scores | as assessed on days 1, 7, 30, 60
  as measured with the visual analog scale (VAS); between 0 and 10; 0 meaning no pain and 10 meaning worst pain possible
Mean Change in Best- Corrected Visual Acuity (BCVA) | from baseline at days 1, 7, 30, 60
  as measured by ETDRS (Early Treatment Diabetic Retinopathy Study) chart
Physician ease of Dextenza insertion | as assessed on day of surgery
  measured by a 0-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Saad Ahmad, MD, Principal Investigator — Kovach Eye Institute
Locations (1):
- Kovach Eye Institute, Elmhurst, Illinois, United States

IPD SHARING:
Plan to Share IPD: No